CLINICAL TRIAL: NCT02768116
Title: A Prospective Multicenter Randomized Trial Comparing Active Transfer of Plaque vs. Provisional T Stenting for the Treatment of Non-Left-Main Coronary Bifurcation Lesions
Brief Title: The Study of Active Transfer of Plaque Technique for Non-Left Main Coronary Bifurcation Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yang Qing, MD, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATP Trial
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Coronary Heart Disease
Keywords: Active Transfer of Plaque
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATP technique (Experimental): This arm plan to enroll 158 subjects. Sirolimus-eluting Drug stent implantation via Active transfer of Plaque technique in the treatment of non-left-main bifurcation lesion.In the ATP technique treatment of bifurcation lesions, by the balloon pre-dilation in the target side branch, the plaque will be actively transferred from side branch to main vessel. Subsequently, the plaque will be fixed by the expansive stent in main vessel. A stent with stent/artery ratio of 1.1:1 is inflated in MV. Rewire to SB is also left at operator's discretion. FKBI or stent in SB is recommended if there is at least one of following: residual stenosis>75%, >type B dissection and TIMI flow<3.
  Interventions: Procedure: Sirolimus Drug-eluting Stent via Active Transfer of Plaque
- Provisional T stenting technique (Active Comparator): This arm plan to enroll 158 subjects. Sirolimus-eluting Drug stent implantation via Provisional T stenting technique in the treatment of non-left-main bifurcation lesions.Provisional T stenting technique is the typic step-T stenting. In brief, two wires are advanced to distal MV and SB. Pre dilation is left at operator's discretion, however, pre dilating SB is not encouraged. Kissing balloon inflation before stenting MV is left at operator's discretion. A stent with stent/artery ratio of 1.1:1 is inflated in MV. Rewire to SB is also left at operator's discretion. FKBI is recommended if there is at least one of following: residual stenosis>75%, >type B dissection and TIMI flow<3.
  Interventions: Procedure: Sirolimus Drug-eluting Stent implantation via Provisional T Stenting

INTERVENTIONS:
Procedure: Sirolimus Drug-eluting Stent via Active Transfer of Plaque
  Arms: ATP technique
Procedure: Sirolimus Drug-eluting Stent implantation via Provisional T Stenting
  Arms: Provisional T stenting technique

SUMMARY:
A Prospective Multi-center Randomized Trial Assessing the Efficacy and Safety of Active Transfer of Plaque vs. Provisional T Stenting for the Treatment of Non-Left-Main Coronary Bifurcation Lesions.

DETAILED DESCRIPTION:
A Prospective Multi-center Randomized Trial Assessing the Efficacy and Safety of Active Transfer of Plaque vs. Provisional T Stenting for the Treatment of Non-Left-Main Coronary Bifurcation Lesions.

The purpose of this trial is to evaluate the efficacy and safety of Active Transfer of Plaque and provisional T stenting techniques treating non-left-main coronary bifurcation lesions based on TLR rate 12-months post-procedure.

Provisional T Stenting is a common technique in BL treatment. Active Transfer of Plaque or ATP was reported, but there are no comparison between two procedure. In the ATP treatment of bifurcation lesions, two wires are advanced to distal main vessel (MV) and side branch(SB). Stent and balloon are advanced to MV and SB respectively. The MV stent is released while dilating the SB balloon. By predilating the balloon in the target SB, the plaque will be actively transferred from SB to MV. Subsequently, the plaque will be fixed by the expansive stent in MV.As to the provisional T treatment, provisional T stenting is the typic step-T stenting. In brief, two wires are advanced to distal MV and SB. Predilation is left at operator's discretion, however, predilating SB is not encouraged. Kissing balloon inflation before stenting MV is left at operator's discretion. A stent with stent/artery ratio of 1.1:1 is inflated in MV. Rewire to SB is also left at operator's discretion. FKBI is recommended if there is at least one of following: residual stenosis>75%, >type B dissection and TIMI flow<3.

All patients will be followed clinically at 1-, 6- 12- and 24-month after stent implantation. Repeat angiographic follow-ups are recommended for all patients at 12 months after the index procedure.

The primary endpoint of the trial is the rate of TLR at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least >18, ≤80 years of age.
* Patient has Stable/unstable angina or NSTEMI.
* Patient has STEMI>24-hour from the onset of chest pain to admission.
* Non-left-main coronary bifurcation lesion. (Medina 0,1,1;1,1,1;1,0,1;1,1,0).
* Patient is eligible for elective percutaneous coronary intervention (PCI) .
* Patient is an acceptable candidate for coronary artery bypass grafting (CABG).
* Patient (or legal guardian) understands the trial requirements and treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed; patient is willing to comply with all protocol-required follow-up evaluations.

Exclusion Criteria:

* Patient with STEMI (within 24-hour from the onset of chest pain to admission).
* Patient has known allergy to the study stent system or protocol-required concomitant medications that cannot be adequately pre-medicated (everolimus, aspirin, contrast media, acrylic acid, Stainless steel).
* Patient has intolerable to dual anti-platelet therapy.
* Patient has any other serious medical illness that may reduce life expectancy to less than 12 months.
* Patient is pregnant or nursing.
* Patient is participating in another clinical trial that has not reached its primary endpoint.
* Patient with severe calcified lesions needing rotational atherectomy.
* Lesions of in-stent restenosis.
* Patients not eligible for this trial based on investigators' judgement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Target lesion revascularization(TLR) rate at 12 months post-procedure | 12 months

SECONDARY OUTCOMES:
Rate of target lesion failure (TLF) at 30days, 6 months, and 24 months, including cardiac death, MI and ischemic TLR. | Up to 2 years
Clinically cardiovascular endpoints at 1-, 6- , 12- and 24-month, including all-cause death, MI and TLR. | Up to 2 years
Stent thrombosis which is defined according to Academic Research Consortium (ARC) definition, including definite, probable and possible stent thrombosis. | Up to 2 years
New York Heart Association classification of cardiac function. | Up to 2 years
Classification score of Canadian Cardiovascular Society (CCS) angina or Braunwald class. | Up to 2 years
In-stent lumen late loss, in-segment and in-stent restenosis rate 12 months after procedure | 12 months

OTHER OUTCOMES:
Procedure success rate | Immediately after procedure
Amount of contrast agent | Immediately after procedure
Procedure time | Immediately after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, MD, PhD, Principal Investigator — Beijing Anzhen Hospital